CLINICAL TRIAL: NCT02770950
Title: Zushima Plaster for Patients in Knee Osteoarthritis: a Random, Positive Drug Controlled, Multi-center Clinical Research
Brief Title: Zushima Plaster for Treating Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Hospital of Traditional Chinese Medicine (Other); Beijing Hospital (Other Government); Beijing Jishuitan Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Gansu Provincial Hospital (Other); General Hospital of Beijing Military Area (Unknown)
Responsible Party: Principal Investigator, Juan Jiao, Attending Doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81758
Record Dates: First submitted 2016-05-02; First posted 2016-05-12 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose group (Active Comparator): High dose of Zushima plaster: a piece of Zushima plaster will be used topically for each knee for 24h per day.
  Eligible subjects will use a piece of Zushima plaster topically for each knee for 24h per day.
  Interventions: Drug: Zushima plaster with high dose
- Low dose group (Active Comparator): Low dose of Zushima plaster: a piece of Zushima plaster will be used topically for each knee for 12h per day.
  Eligible subjects will use a piece of Zushima plaster topically for each knee for 12h per day.
  Interventions: Drug: Zushima plaster with low dose
- Controlled group (Active Comparator): Indometacin Cataplasms will be used topically on the knee for 24h per day
  Interventions: Drug: Indometacin Cataplasms

INTERVENTIONS:
Drug: Zushima plaster with high dose — Patients in high dose Zushima plaster group will use Zushima plaster topically on knee(s) for 24h per day.
  Arms: High dose group
Drug: Zushima plaster with low dose — Patients in low dose Zushima plaster group will use Zushima plaster topically on knee(s) for 12h per day.
  Arms: Low dose group
Drug: Indometacin Cataplasms — Patients in Indometacin Cataplasms group will use Indometacin Cataplasms on knee(s)for 24h per day.
  Arms: Controlled group

SUMMARY:
The purpose of this study is to further evaluate the clinical efficacy and safety of Zushima plaster for patients in knee osteoarthrosis post-marketing.

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-75;
* Unilateral or bilateral knee OA, confirmed radiographically;
* Patients taking oral NSAIDs prior to the breakthrough period will be permitted;
* VAS pain score is or above 20mm.

Exclusion Criteria:

* Knee is swollen and hot;
* Allergic to any ingredient in Girald Daphne Bark Plaster (Girald Daphne Bark, Lithargite, Linseed oil, Red lead) ;
* Congestive Heart Failure and Edema;
* Advanced renal disease;
* Knee joint skin is burst or skin disease or allergies.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the change of Visual Analogue Scale (VAS) pain score from baseline to posttreatment | Week 2.

SECONDARY OUTCOMES:
the change of Patient's global assessment of disease activity from baseline to posttreatment | Week 2.
the change of WOMAC Osteoarthritis Index from baseline to posttreatment | Week 2.
the change of Short Form 36 Questionnaire (SF-36) score from baseline to posttreatment | Week 2.
  The SF-36 is a generic instrument to assess health-related quality of life. It consists of 36 questions and assesses 8 dimensions: physical functioning, role physical, pain index, general health, vitality, social functioning, role emotional, and mental health index. It also provides 2 summary measures of physical and mental components. The SF-36 score ranges from 0 to 100, with higher scores indicating better health status.
the change of Erythrocyte Sedimentation rate (ESR) from baseline to posttreatment | Week 2.
  ESR, also called a sedimentation rate, is the rate at which red blood cells sediment in a period of one hour. It is a non-specific measure of inflammation.
the change of C-reactive protein (CRP) from baseline to posttreatment | Week 2.
the change of knee musculoskeletal ultrasound (MSUS) from baseline to posttreatment | Week 2.
  MSUS had wisely using in rheumatology practice and research. MSUS includes synovitis classification, synovial hyperplasia classification, articular cavity effusion and bone erosion classification. Specific as follows: Synovitis classification: 0 level, no doppler signal; level 1: three independent point or 2 successive or 1 and 2 in independent dot doppler signal; level 2: doppler signal < 50% of the synovial membrane area; level 3 doppler signal is the synovium in > 50% of the area. Synovial hyperplasia classification: 0 level, no synovial hyperplasia; level 1: synovial hyperplasia of mild, not more than bone surface high attachment; level 2: synovial hyperplasia more than bone surface high wire, but not more than the backbone; level 3: synovial hyperplasia more than bone surface peak wires, and extends along the backbone of the side. Articular cavity effusion and bone erosion classification: adopt binary evaluation, namely 0: normal, 1: abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Jiang, MD. PhD., Principal Investigator — Rheumatology Department
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided